CLINICAL TRIAL: NCT00886691
Title: A Phase II Randomized, Double-Blinded Evaluation of Oral Everolimus (RAD001) Plus Bevacizumab vs. Oral Placebo Plus Bevacizumab in the Treatment of Recurrent or Persistent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Bevacizumab With or Without Everolimus in Treating Patients With Recurrent or Persistent Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GOG Foundation (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GOG-0186G; NCI-2011-01914 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000640439; GOG-0186G (Other: NRG Oncology); GOG-0186G (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2018-07-02 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Everolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (bevacizumab and everolimus) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and everolimus PO QD on days 1-28.
  Interventions: Biological: Bevacizumab; Drug: Everolimus; Other: Laboratory Biomarker Analysis
- Arm II (bevacizumab and placebo) (Experimental): Patients receive bevacizumab as in Arm I and placebo PO QD on days 1-28.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Other: Placebo

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; BEVACIZUMAB, LICENSE HOLDER UNSPECIFIED; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
  Arms: Arm I (bevacizumab and everolimus)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (bevacizumab and placebo)

SUMMARY:
This randomized phase II trial studies how well bevacizumab with or without everolimus works in treating patients with recurrent or persistent ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Bevacizumab and everolimus may also stop the growth of tumor cells by blocking blood flow to the tumor. It is not yet known whether bevacizumab is more effective when given together with or without everolimus in treating ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the progression-free survival hazard ratio of the combination of oral everolimus (RAD001) and bevacizumab compared to oral placebo and bevacizumab in patients with persistent or recurrent ovarian, fallopian tube, or primary peritoneal cancer.

SECONDARY OBJECTIVES:

I. To determine the nature and degree of toxicity of oral everolimus (or placebo) plus bevacizumab.

II. To characterize and compare progression-free survival and overall survival in patients with measurable disease (Response Evaluation Criteria in Solid Tumors [RECIST] criteria) and patients with detectable (non-measurable) disease.

III. To estimate the proportion of patients with measurable disease who have objective tumor responses by treatment.

IV. To provide descriptive information about cancer antigen (CA)-125 responses by regimen and where possible by objective tumor responses.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive bevacizumab intravenously (IV) over 30-90 minutes on days 1 and 15 and everolimus orally (PO) once daily (QD) on days 1-28.

ARM II: Patients receive bevacizumab as in Arm I and placebo PO QD on days 1-28.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma; histologic documentation of the original primary tumor is required via the pathology report
* Patients must have measurable disease or detectable (non-measurable) disease:

  * Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each lesion must be greater than or equal to 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or greater than or equal to 20 mm when measured by chest x-ray; lymph nodes must be greater than or equal to 15 mm in short axis when measured by CT or MRI
  * Detectable disease in a patient is defined as one who does not have measurable disease but has at least one of the following conditions:

    * Baseline values of CA-125 at least 2 x upper limit of normal (ULN)
    * Ascites and/or pleural effusion attributed to tumor
    * Solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions
* Patients in the measurable disease cohort must have at least one ?target lesion? to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as ?non-target? lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG phase III protocol or Rare Tumor Protocol for the same patient population
* Patients who have had one prior treatment must have a GOG performance status of 0, 1, or 2; patients who have had two or three prior treatments must have a GOG performance status of 0 or 1
* Patients should be free of active infection requiring parenteral antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy

  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
  * Any other prior therapy directed at the malignant tumor, including biological and immunologic agents, must be discontinued at least 3 weeks prior to registration (including small molecules and murine monoclonal antibodies); chimeric or human or humanized monoclonal antibodies (including bevacizumab) or vascular endothelial growth factor (VEGF) receptor fusion protein (including VEGF Trap, aflibercept) must be discontinued for at least 12 weeks prior to registration; no investigational therapy within 30 days prior to the first date of study treatment
* Prior therapy:

  * Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound' this initial treatment may have included intraperitoneal therapy, consolidation, non-cytotoxic agents or extended therapy administered after surgical or non-surgical assessment
  * Patients are allowed to receive, but are not required to receive, two additional cytotoxic regimens for management of recurrent or persistent disease, with no more than 1 non-platinum, non-taxane regimen
  * Patients are allowed to receive, but are not required to receive, biologic (non-cytotoxic) therapy as part of their primary treatment regimen; patients must have NOT received any non-cytotoxic therapy for management of recurrent or persistent disease
  * Patients who have received only one prior cytotoxic regimen (platinum-based regimen for management of primary disease), must have a platinum-free interval of less than 12 months, or have progressed during platinum-based therapy, or have persistent disease after a platinum-based therapy
  * For the purposes of this study, poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitors will be considered ?cytotoxic,? and prior treatment with PARP inhibitors for primary or recurrent disease WILL be allowed (either alone or in combination with chemotherapy)
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl
* Platelets greater than or equal to 100,000/mcl
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN)
* Bilirubin less than or equal to 1.5 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) less than or equal to 3 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Prothrombin time (PT) such that international normalized ratio (INR) is less than or equal to 1.5 x ULN (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin for management of deep vein thrombosis including pulmonary embolism)
* Partial thromboplastin time (PTT) less than or equal to 1.5 times the upper limit of normal
* Fasting serum cholesterol less than or equal to 300 mg/dL OR less than or equal to 7.75 mmol/L AND
* Fasting triglycerides less than or equal to 300 mg/dL or 3.42 mmol/L
* Urine protein creatinine (UPC) ratio must be < 1.0 gm; if UPC ratio >= 1, collection of 24-hour urine measurement of urine protein is recommended; UPC ratio of spot urine is an estimation of the 24-hour urine protein excretion?a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 gm
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing an effective form of contraception
* Patients must have signed an approved informed consent and authorization permitting the release of personal health information
* Patients must meet pre-entry requirements
* Patients with clinically significant cardiovascular disease; this includes:

  * Uncontrolled hypertension, defined as systolic > 150 mm Hg or diastolic > 90 mm Hg
  * Myocardial infarction or unstable angina within 6 months prior to registration
  * New York Heart Association (NYHA) class II or greater congestive heart failure
  * Serious cardiac arrhythmia requiring medication; this does not include asymptomatic, atrial fibrillation with controlled ventricular rate
  * Patients who have received prior treatment with an anthracycline (including doxorubicin and or liposomal doxorubicin) and have an ejection fraction < 50%
  * Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or greater peripheral vascular disease (at least brief [< 24 hours (hrs)] episodes of ischemia managed non-surgically and without permanent deficit)

Exclusion Criteria:

* Patients who have received prior everolimus or any other mammalian target of rapamycin (mTOR) inhibitor
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies, are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of ovarian, fallopian tube or primary peritoneal cancer within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian, fallopian tube or primary peritoneal cancer within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients with serious non-healing wound, ulcer, or bone fracture; this includes history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days prior to the first date of study treatment
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months prior to the first date of study treatment
* Known hypersensitivity to murine or chimeric antibodies
* Major surgery within 28 days prior to the first date of study treatment
* Patients with clinical symptoms or signs of gastrointestinal obstruction and patients who require parenteral hydration and/or nutrition
* Patients with medical history or conditions not otherwise previously specified which in the opinion of the investigator should exclude participation in this study; the investigator can consult the Study Chair or Study Co-Chairs for uncertainty in this regard
* Patients who are pregnant or nursing
* Patients with active hepatitis B or C

  * Laboratory confirmation to exclude hepatitis B and C is required in any patient considered at high risk for hepatitis B or C; risk factors can include:

    * You currently live in (or have lived in) Asia, Africa, Central and South America, Eastern Europe, Spain, Portugal, and Greece
    * Known or suspected past hepatitis B infection
    * Known or suspected past hepatitis C infection (including past interferon ?curative? treatment)
    * Blood transfusion(s) prior to 1990
    * Current or prior IV drug use
    * Current or prior dialysis
    * Household contact with hepatitis B or hepatitis C infected person(s)
    * Current or prior high-risk sexual activity
    * Body piercing or tattoos
    * Mother known to have hepatitis B
    * History suggestive of hepatitis B infection, e.g., dark urine, jaundice, right upper quadrant pain

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-12-27 (Actual); Primary Completion 2014-06-27 (Actual); Study Completion 2015-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William P Tew, Principal Investigator — NRG Oncology
Locations (45):
- United States (45):
  - Gynecologic Oncology Group of Arizona, Phoenix, Arizona
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Hospital, Aurora, Colorado
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Rush University Medical Center, Chicago, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Baystate Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - LDS Hospital, Salt Lake City, Utah
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 150 patients were enrolled into this trial. The study opened to accrual December 2010 and closed to patient entry August 2012.
Groups:
- Everolimus (RAD001) Plus Bevacizumab: EVEROLIMUS (RAD001) 10mg orally daily plus Bevacizumab IV at 10 mg/kg Day 1 and Day 15 (one cycle = 4 weeks)
- Placebo Plus Bevacizumab: ORAL PLACEBO daily plus Bevacizumab IV at 10 mg/kg Day 1 and Day 15 (one cycle = 4 weeks)
Period: Overall Study
Arm/Group | Everolimus (RAD001) Plus Bevacizumab | Placebo Plus Bevacizumab
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All intent to treat patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus (RAD001) Plus Bevacizumab | Placebo Plus Bevacizumab | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 1 | 0 | 1
  30-39 years | 1 | 1 | 2
  40-49 years | 9 | 8 | 17
  50-59 years | 16 | 21 | 37
  60-69 years | 33 | 28 | 61
  70-79 years | 12 | 13 | 25
  >=80 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 75 | 150
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: The time from randomization until disease progression, death, or date of last contact. Endpoints are progression or death. Patients who are not observed with an endpoint are censored. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) as an 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Duration of time from start of treatment to time of progression, approximately 4 years and 6 months.
Population: All intent to treat patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus (RAD001) Plus Bevacizumab | Placebo Plus Bevacizumab
Number analyzed (Participants) | 75 | 75
months | 5.9 [4.11 to 7.69] | 4.5 [3.75 to 6.90]

2. Secondary Outcome: Incidence of Adverse Events as Assessed by Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.0)
Description: Number of participants with a grade of 3 or higher during the treatment period.
Time Frame: All Adverse Events (AEs) and Serious Adverse Events (SAEs) occurring during treatment and up to 30 days after stopping the study treatment, approximately 4 years and 6 months.
Population: All Intent to treat patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus (RAD001) Plus Bevacizumab | Placebo Plus Bevacizumab
Number analyzed (Participants) | 75 | 75
Participants | 43 | 20

3. Secondary Outcome: Characterize and Compare Progression-free Survival and Overall Survival in Patients With Measurable Disease (RECIST Criteria) and Patients With Detectable (Non-measurable) Disease
Description: Progression-free survival and overall survival broken down by measurable disease status
Time Frame: Continued until disease progression, assessed up to approximately 4 years and 6 months
Population: All Intent to treat patients
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- PFS (Progression Free Survival) in Non-measurable Patients; OS (Overall Survival) in Non-measurable Patients: Patients with non- measurable disease
- PFS (Progression Free Survival) in Measurable Patients; OS (Overall Survival) in Measurable Patients: Patients with measurable disease
Arm/Group | PFS (Progression Free Survival) in Non-measurable Patients | PFS (Progression Free Survival) in Measurable Patients | OS (Overall Survival) in Non-measurable Patients | OS (Overall Survival) in Measurable Patients
Number analyzed (Participants) | 29 | 121 | 29 | 121
Months | 3.94 [2.63 to 5.82] | 5.91 [4.27 to 7.43] | 11.10 [7.59 to NA] — Insufficient follow-up time | 16.92 [12.16 to 18.43]

4. Secondary Outcome: The Proportion of Patients With Measurable Disease Who Have Objective Tumor Responses by Treatment.
Description: Complete and Partial Tumor Response by RECIST 1.0
Time Frame: Up to approximately 4 years and 6 months
Population: All measurable patients treated on Everolimus plus Bevicizumab and Placebo plus Bevacizumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants responding
Arm/Group | Everolimus (RAD001) Plus Bevacizumab | Placebo Plus Bevacizumab
Number analyzed (Participants) | 63 | 58
percentage of participants responding | 22.2 [12.7 to 34.5] | 12.1 [5.0 to 23.3]

5. Secondary Outcome: Percentage of Participants With at Least One Cancer Antigen 125 (CA-125) Response
Description: Response as evaluated by CA-125 levels.A CA 125 test measures the amount of the protein CA 125 (cancer antigen 125) in blood.CA 125 is a tumor marker recommended for clinical use in the diagnosis and management of ovarian cancer. CA-125 responses were assessed with Rustin criteria. Initial values had to be 2x ULN (upper limit of normal) within 2 weeks of starting therapy to be considered evaluable.Patient were evaluated by using best overall response while receiving study therapy.
Time Frame: Prior to each cycle of treatment. Then follow-up every three months for 2 years , then every 6 months for 3 years. Duration was approximately 4 years and 6 months.
Population: CA-125 evaluable patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Everolimus (RAD001) Plus Bevacizumab | Placebo Plus Bevacizumab
Number analyzed (Participants) | 44 | 39
percentage of participants | 27.3 [15.0 to 42.8] | 15.4 [5.9 to 30.5]

ADVERSE EVENTS:
Time Frame: Study Treatment and up to 30 days after stopping study treatment, up to approximately 4 years and 6 months.
Description: The frequencies of any serious adverse event or other adverse events by category or specific term occurring during treatment and up to 30 days after stopping the study treatment are reported.
Arm/Group | Everolimus (RAD001) Plus Bevacizumab | Placebo Plus Bevacizumab
Serious Adverse Events (participants affected / at risk) | 35/75 | 24/75
Other Adverse Events (participants affected / at risk) | 73/75 | 72/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (RAD001) Plus Bevacizumab (N=75) | Placebo Plus Bevacizumab (N=75)
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Colonic Obstruction (Gastrointestinal disorders) | 1 | 1
Colonic Perforation (Gastrointestinal disorders) | 3 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 2
Abdominal Pain (Gastrointestinal disorders) | 3 | 1
Obstruction Gastric (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Ascites (Gastrointestinal disorders) | 2 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Death Nos (General disorders) | 1 | 1
Fever (General disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 2 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1
Catheter Related Infection (Infections and infestations) | 0 | 1
Anorectal Infection (Infections and infestations) | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Lymphocyte Count Decreased (Investigations) | 1 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal And Connective Tissue Disorder - (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Treatment Related Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intracranial Hemorrhage (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thromboembolic Event (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 1 | 1
Hematoma (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (RAD001) Plus Bevacizumab (N=75) | Placebo Plus Bevacizumab (N=75)
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 52 | 26
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 4 | 3
Heart Failure (Cardiac disorders) | 1 | 0
Atrial Flutter (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 4 | 0
Chest Pain - Cardiac (Cardiac disorders) | 1 | 0
Ear And Labyrinth Disorders - Other (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Hearing Impaired (Ear and labyrinth disorders) | 2 | 2
Ear Pain (Ear and labyrinth disorders) | 4 | 0
External Ear Pain (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Endocrine Disorders - Other (Endocrine disorders) | 1 | 0
Eye Disorders - Other (Eye disorders) | 1 | 0
Watering Eyes (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 1
Blurred Vision (Eye disorders) | 7 | 5
Dry Eye (Eye disorders) | 0 | 1
Floaters (Eye disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 9 | 1
Dyspepsia (Gastrointestinal disorders) | 10 | 7
Duodenal Obstruction (Gastrointestinal disorders) | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 1 | 1
Colonic Obstruction (Gastrointestinal disorders) | 0 | 1
Colonic Perforation (Gastrointestinal disorders) | 1 | 0
Colonic Fistula (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 33 | 26
Diarrhea (Gastrointestinal disorders) | 36 | 28
Vomiting (Gastrointestinal disorders) | 31 | 19
Bloating (Gastrointestinal disorders) | 14 | 6
Small Intestinal Perforation (Gastrointestinal disorders) | 1 | 0
Stomach Pain (Gastrointestinal disorders) | 1 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1
Anal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Anal Mucositis (Gastrointestinal disorders) | 1 | 0
Rectal Fistula (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 25 | 22
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal Hemorrhage (Gastrointestinal disorders) | 2 | 1
Oral Dysesthesia (Gastrointestinal disorders) | 1 | 0
Obstruction Gastric (Gastrointestinal disorders) | 0 | 1
Mucositis Oral (Gastrointestinal disorders) | 44 | 14
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Anal Pain (Gastrointestinal disorders) | 0 | 1
Oral Hemorrhage (Gastrointestinal disorders) | 1 | 2
Ileus (Gastrointestinal disorders) | 1 | 0
Anal Ulcer (Gastrointestinal disorders) | 0 | 1
Gingival Pain (Gastrointestinal disorders) | 2 | 0
Oral Pain (Gastrointestinal disorders) | 4 | 2
Abdominal Distension (Gastrointestinal disorders) | 11 | 5
Nausea (Gastrointestinal disorders) | 39 | 33
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 3
Rectal Pain (Gastrointestinal disorders) | 2 | 0
Lip Pain (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 2 | 0
Hemorrhoids (Gastrointestinal disorders) | 7 | 1
Ascites (Gastrointestinal disorders) | 2 | 3
Toothache (Gastrointestinal disorders) | 3 | 1
Dental Caries (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Pain (General disorders) | 14 | 7
Malaise (General disorders) | 2 | 0
Irritability (General disorders) | 0 | 2
Flu Like Symptoms (General disorders) | 3 | 0
Edema Trunk (General disorders) | 2 | 1
Non-Cardiac Chest Pain (General disorders) | 3 | 2
Edema Limbs (General disorders) | 7 | 5
Edema Face (General disorders) | 2 | 0
Fatigue (General disorders) | 61 | 56
Fever (General disorders) | 11 | 6
Gait Disturbance (General disorders) | 0 | 1
Chills (General disorders) | 9 | 3
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Allergic Reaction (Immune system disorders) | 2 | 0
Infections And Infestations - Other (Infections and infestations) | 2 | 0
Upper Respiratory Infection (Infections and infestations) | 2 | 3
Tooth Infection (Infections and infestations) | 3 | 2
Skin Infection (Infections and infestations) | 6 | 1
Sinusitis (Infections and infestations) | 6 | 3
Sepsis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Otitis Media (Infections and infestations) | 1 | 1
Otitis Externa (Infections and infestations) | 1 | 0
Nail Infection (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 1 | 1
Laryngitis (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Device Related Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 11 | 3
Lip Infection (Infections and infestations) | 0 | 1
Anorectal Infection (Infections and infestations) | 1 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Burn (Injury, poisoning and procedural complications) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 3 | 1
Weight Loss (Investigations) | 15 | 9
Weight Gain (Investigations) | 1 | 2
Serum Amylase Increased (Investigations) | 0 | 1
Platelet Count Decreased (Investigations) | 39 | 9
Lymphocyte Count Decreased (Investigations) | 7 | 5
Lipase Increased (Investigations) | 0 | 1
Inr Increased (Investigations) | 4 | 1
Ggt Increased (Investigations) | 0 | 1
Creatinine Increased (Investigations) | 11 | 4
Cholesterol High (Investigations) | 29 | 11
Neutrophil Count Decreased (Investigations) | 33 | 7
Cardiac Troponin I Increased (Investigations) | 1 | 0
Cpk Increased (Investigations) | 1 | 0
Blood Bilirubin Increased (Investigations) | 1 | 2
White Blood Cell Decreased (Investigations) | 34 | 11
Aspartate Aminotransferase Increased (Investigations) | 22 | 3
Alkaline Phosphatase Increased (Investigations) | 16 | 6
Alanine Aminotransferase Increased (Investigations) | 15 | 6
Activated Partial Thromboplastin Time Prolonged (Investigations) | 2 | 0
Metabolism And Nutrition Disorders - Other (Metabolism and nutrition disorders) | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 10 | 1
Hyponatremia (Metabolism and nutrition disorders) | 14 | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 15 | 9
Hypokalemia (Metabolism and nutrition disorders) | 18 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 17 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 20 | 7
Hyperuricemia (Metabolism and nutrition disorders) | 6 | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 24 | 8
Hypernatremia (Metabolism and nutrition disorders) | 4 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 27 | 11
Glucose Intolerance (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 1
Anorexia (Metabolism and nutrition disorders) | 34 | 15
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 10 | 5
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 18
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 3 | 0
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 5 | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Buttock Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 16
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 20
Musculoskeletal And Connective Tissue Disorder - (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tremor (Nervous system disorders) | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 25 | 25
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 2
Paresthesia (Nervous system disorders) | 2 | 3
Memory Impairment (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 31 | 29
Dysphasia (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 9 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 9 | 8
Cognitive Disturbance (Nervous system disorders) | 2 | 0
Psychiatric Disorders - Other (Psychiatric disorders) | 0 | 1
Libido Decreased (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 15 | 9
Hallucinations (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 8 | 12
Confusion (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 12 | 8
Agitation (Psychiatric disorders) | 0 | 1
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 1 | 0
Urine Discoloration (Renal and urinary disorders) | 1 | 0
Urinary Urgency (Renal and urinary disorders) | 3 | 0
Urinary Retention (Renal and urinary disorders) | 2 | 1
Urinary Incontinence (Renal and urinary disorders) | 1 | 1
Urinary Tract Pain (Renal and urinary disorders) | 5 | 0
Urinary Frequency (Renal and urinary disorders) | 8 | 1
Proteinuria (Renal and urinary disorders) | 6 | 6
Hemoglobinuria (Renal and urinary disorders) | 2 | 1
Hematuria (Renal and urinary disorders) | 2 | 0
Cystitis Noninfective (Renal and urinary disorders) | 1 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 0
Bladder Spasm (Renal and urinary disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 0
Vaginal Pain (Reproductive system and breast disorders) | 1 | 0
Vaginal Hemorrhage (Reproductive system and breast disorders) | 0 | 4
Vaginal Dryness (Reproductive system and breast disorders) | 1 | 1
Pelvic Pain (Reproductive system and breast disorders) | 4 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 3 | 3
Vaginal Inflammation (Reproductive system and breast disorders) | 1 | 0
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 10 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pharyngeal Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 26 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 18
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 7 | 5
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 3
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 2 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 17 | 3
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Nail Ridging (Skin and subcutaneous tissue disorders) | 1 | 2
Nail Loss (Skin and subcutaneous tissue disorders) | 2 | 2
Nail Discoloration (Skin and subcutaneous tissue disorders) | 5 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 10
Surgical And Medical Procedures - Other (Surgical and medical procedures) | 1 | 0
Thromboembolic Event (Vascular disorders) | 2 | 4
Lymphedema (Vascular disorders) | 2 | 3
Hypertension (Vascular disorders) | 24 | 31
Hot Flashes (Vascular disorders) | 5 | 9
Hematoma (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less